CLINICAL TRIAL: NCT02565017
Title: Examining Patient Preferences About the IBM Watson Oncology Clinical Decision Support System
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-226
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer
Keywords: IBM Watson; Clinical Decision Support System; Patient Preferences; 15-226
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Patient Preference | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Breast Cancer: and treatment type (chemotherapeutic adjuvant (i.e., chemotherapy delivered after primary therapy/surgery) or neoadjuvant (i.e., chemotherapy delivered prior to primary therapy/surgery) treatment, chemotherapeutic treatment for metastatic disease, or chemotherapeutic treatment through a clinical trial).
  Interventions: Behavioral: Focus groups
- Lung Cancer: and treatment type (chemotherapeutic adjuvant (i.e., chemotherapy delivered after primary therapy/surgery) or neoadjuvant (i.e., chemotherapy delivered prior to primary therapy/surgery) treatment, chemotherapeutic treatment for metastatic disease, or chemotherapeutic treatment through a clinical trial).
  Interventions: Behavioral: Focus groups
- Colorectal Cancer: and treatment type (chemotherapeutic adjuvant (i.e., chemotherapy delivered after primary therapy/surgery) or neoadjuvant (i.e., chemotherapy delivered prior to primary therapy/surgery) treatment, chemotherapeutic treatment for metastatic disease, or chemotherapeutic treatment through a clinical trial).
  Interventions: Behavioral: Focus groups

INTERVENTIONS:
Behavioral: Focus groups — After the presentation of the of IBM Watson Oncology at the opening of the focus group, participants will be asked to fill out a de-identified brief 15-item questionnaire to assess participants' first impressions of IBM Watson Oncology. The questionnaire will be self administered, and will take approximately 5 minutes to complete. Completed questionnaires will be collected by a member of the study staff, and the focus group will proceed with introductions. The focus group will be audio recorded from the completion of the introductions and notes will be taken. The focus group guide will address the study aims. At the end of the focus group, participants will complete a 7-item questionnaire to capture simple demographic information including education, income, and health literacy. This questionnaire will take 3-5 minutes to complete.

SUMMARY:
The purpose of this study is to learn what cancer patients think about IBM Watson Oncology. IBM Watson Oncology is a computer program designed to help inform oncologists about the best chemotherapy choices for their patients. The investigators will conduct focus groups with cancer patients who have received chemotherapy treatment at MSK in order to understand cancer patients' thoughts about IBM Watson Oncology.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC patient 18 years or older
* Breast, lung, or colorectal cancer MSK patient as per EMR or clinician judgment having either:

  * Chemotherapeutic adjuvant or neoadjuvant treatment with the first chemo visit occurring within the past 8 months and primary treatment (i.e., surgery), occurring within the past 6 months)at MSK
  * OR chemotherapeutic treatment for metastatic disease with the first chemo visit occurring within the past 8 months at MSK
  * OR chemotherapeutic treatment through an on-going MSK clinical trial as per clinician
* Residing in New York metro-area

Exclusion Criteria:

* Non-English speakers because we do not have the resources to conduct and translate the focus groups into other languages
* Patients who are not or will not receive their cancer care at MSKCC.
* Patient unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Acceptability of IBM Watson Oncology | 1 year
  Data collected through the brief questionnaires (e.g.,initial impressions of IBM Watson Oncology, sociodemographics) will be entered into an SPSS data file on the secure MSK server.

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamilton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/